CLINICAL TRIAL: NCT06459700
Title: Effect of 6 Months Probiotic Supplement on Pain, Function, Quality of Life and Inflammation in Females With Knee Osteoarthritis: A Double-blinded Randomized Placebo-controlled Trial
Brief Title: Effect of Probiotic Supplements on Osteoarthritis Outcomes
Acronym: ProOA23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ProOA23
Record Dates: First submitted 2024-05-22; First posted 2024-06-14 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): One arm will receive probiotic supplement in opaque white capsules, 1 each day for six months
  Interventions: Dietary Supplement: Probiotic supplements
- Placebo (Placebo Comparator): One arm will receive identical opaque placebo capsules containing maize starch powder (placebo), 1 each day for six months
  Interventions: Dietary Supplement: Placebo supplements

INTERVENTIONS:
Dietary Supplement: Probiotic supplements — See arm/group description
  Arms: Probiotic
Dietary Supplement: Placebo supplements — See arm/group description
  Arms: Placebo

SUMMARY:
Dysbiosis of the gut microbiota is believed to contribute to the development and progression of osteoarthritis (OA), suggesting a role for probiotics in the treatment of OA. Animal studies have shown that certain probiotic strains decrease the inflammatory responses, pain sensitization and OA progression. There are, however, few clinical studies in humans to support this. In this double-blinded randomized controlled trial we will investigate the effect of 6-months probiotic supplements compared to placebo on OA related outcomes in females with diagnosed knee OA.

DETAILED DESCRIPTION:
Aim:

To investigate the effect of 6-moths probiotic supplements compared to placebo on OA related outcomes in females with diagnosed knee OA.

Design: Double-blinded randomized placebo controlled trial

Study arms: One treatment arm will receive probiotic supplement in opaque white capsules and the other treatment arm will receive identical opaque placebo capsules. The placebo product will contain maize starch powder. Study participants will take one capsule daily for six months.

Statistical analysis Main outcome: The independent T-test will be used to evaluate group differences in change in KOOS-12 scores between baseline and 6-months follow-up, given that all assumptions for parametric tests are satisfied. If assumptions are not met or if there are differences in baseline characteristics due to imbalanced randomization the Mann-Whitney U-test or regression analysis will be used as appropriate.

Secondary and explorative outcomes: The independent T-test (continuous, normal distributed data), the Mann-Whitney U-test (ordinal, non-normally distributed data) and cross-tabulations with Chi2 test (nominal data) will be used to evaluate differences in secondary and explorative outcomes between the two groups.

Estimated enrollment: 86 participants. Based on the ability to detect a 10-score difference in KOOS-12 with 80% power and α 0.05, 72 participants (36 per arm) will be needed. With an approximate drop-out rate of 20% from baseline to follow-up, 86 participants will be recruited.

Investigators: Eva Ageberg, PT, PhD, Professor in physical therapy, Lund University, Sweden (Principal investigator), Anna Cronström, physical therapist, PhD, Lund University, Sweden, Jessica Neilands, PhD, Associate Professor, Science manager, Probi AB, Lund, Sweden and Daniel Benoit, PhD, senior lecturer in Experimental Health Sciences at Lund University, Sweden.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 45-70 years
2. Clinical diagnosis of knee OA
3. Mild to moderate knee joint pain (Visual Analog Scale (VAS) 3-7)) during the last 3 months
4. Able to perform walking and stair tests
5. No use of other supplements/food products containing probiotics and/or supplements targeting OA symptoms (e.g., glucosamine, turmeric)
6. Able to write and understand Swedish.

Exclusion Criteria:

1. Rheumatoid arthritis or other active generalised inflammatory comorbidities affecting the gastrointestinal tract (IBD, celiac disease)
2. Performed a total knee replacement on the affected knee or on waiting list for joint replacement
3. Other concomitant injuries or surgeries overriding the OA knee symptoms
4. Other concomitant injuries or diseases where physical activity is a contra indication
5. Malabsorption disorders, presence of renal and/or hepatic failure
6. Use of corticosteroids with doses above 10 mg/day and/or Intra-articular injections during the previous 6 months
7. Heavy use of alcohol (>10 standard units a week), or recreational drug use
8. BMI ≥30 Kg/m2
9. Antibiotic treatment during the previous 2 months
10. clinical depression diagnosis
11. Pregnancy/breast feeding
12. Smoking or other nicotine containing products during the previous 6months
13. Performed a gastric bypass
14. Immunosuppressive treatment or impaired immune system
15. Chronic or acute diarrhoea
16. Blood/plasma donation/transfusion during the 3months or during the study
17. Non-controlled diabetes
18. Allergy with regards to any of the study product ingredients.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS)-12 | 6 months
  Change in the KOOS-12 (total score) from baseline to 6 months in the probiotic group compared with the placebo group. The KOOS-12 is scored from 1-100 (worst-best) scale.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (separate subscale score) | 3 to 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline to 3-month and 6-month follow-up in Scores on the separate subscales (pain, symptoms, activity of daily living, sport/recreation and knee-related quality of life) from the full KOOS questionnaire. The KOOS is scored from 1-100 (worst-best) scale.
Visual Analogue Scale (VAS) | 3 to 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline to 3-month and 6-month follow-up in VAS scores (pain severity), assessed on an ordinal scale from 0 to 10 where 0 indicates no pain and 10 worst possible pain the last week
Work Productivity and Activity Impairment questionnaire (WPAI) | 3 to 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline to 3-month and 6-month follow-up in WPAI. The WPAI questionnaire includes 6 questions regarding employee's absenteeism, reduced job performance, work productivity loss, and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Patient Acceptable Symptom State (PASS) | 3 to 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline to 3-month and 6-month follow-up in PASS. The PASS involves a question regarding if the patient is satisfied with their current knee function with to response options (yes/no)
Pain-relieving medication intake | 3 to 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline to 3-month and 6-month follow-up in pain-relieving medication intake. Here the patients reports the type and dosage of any medication
Wish for surgery | 3 to 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline to 3-month and 6-month follow-up in wish for surgery. The patients are asked if they wish to undergo surgery due to their knee problems (yes/no).
40m fast paced walk test | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in 40m fast paced walk test, assessed as time taken to walk 4x10 meter as fast as possible
30 seconds sit to stand test | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in the 30 seconds sit to stand test, assessed by the number of repetitions of sitting to standing from a chair during a period of 30 second.
Stair climb test | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in the stair climb test, assessed as time taken to ascend and descend a flight of 5 stairs.
3 minute walk test | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in the 3 minute walk test, assessed as distance walked during 3 minutes on a treadmill.
Molecular biomarkers for cartilage degeneration and inflammation. | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in molecular biomarkers for cartilage degeneration and inflammation.

OTHER OUTCOMES:
Kinematics assessed with 3D motion analysis | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in Kinematics (joint angles in degrees) during the functional tasks
Kinetics assessed with 3D motion analysis and force plates | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up in kinetics (joint moments (newton meter)) during the functional tasks.
Intestinal barrier integrity | 6 months
  Comparison of the probiotic group with the placebo group in terms of changes from baseline and 6-month follow-up a molecular biomarker for intestinal barrier integrity (Zonulin)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, Principal Investigator — Lund University
Locations (1):
- MoReLab, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Plan description: De-identified IPD for primary and secondary outcomes will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Statistical analysis plan will be published in a study protocol before completion of the analysis.